CLINICAL TRIAL: NCT02431494
Title: Safety and Preliminary Efficacy of Combination Blue Light Phototherapy and Microcurrent Therapy for the Treatment of Acne Vulgaris
Brief Title: Safety and Preliminary Efficacy of Combination Therapy for the Treatment of Acne Vulgaris
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Nova Southeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08291420Exp
Record Dates: First submitted 2015-04-21; First posted 2015-05-01 (Estimated); Results first posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Acne Vulgaris; Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BLP arm (Blue Light Phototherapy) (Active Comparator): In this arm participants will receive 5 BLP sessions at 1 week intervals. The duration of each session will be approximately 20 minutes. At each session, the affected areas of the participant's face will be exposed to a light source using blue light phototherapy machine between 15 to 20 minutes.
  Interventions: Device: Blue light phototherapy
- MCT arm (Microcurrent Therapy) (Active Comparator): In this arm participants will receive 5 MCT sessions 1 week intervals using MCT machine. The duration of each session will be approximately 45 minutes. The investigators will place one electrode in one of the regional areas of the lymph nodes or affected area (i.e. the forehead) and move the second electrode systematically from the affected area towards the stationary electrode. Once the entire affected area has been covered, the investigators will move the first electrode to another regional area of the lymph nodes or affected area and the process will be repeated. This will continue until all of the affected areas have been treated.
  Interventions: Device: Microcurrent therapy
- Combination of BLP and Microcurrent (Active Comparator): In this arm participants will receive 5 BLP and 5 MCT sessions at 1 week intervals. At each session, participants will receive MCT portion as described in above followed by BLP portion as described above. These visits will last approximately 65 minutes.
  Interventions: Device: Combination of BLP and Microcurrent

INTERVENTIONS:
Device: Blue light phototherapy — Blue light phototherapy (BLU-U Blue Light Photodynamic Therapy Illuminator manufactured by DUSA Pharmaceutical Inc. Wilmington, MA) At each session, the affected areas of the participant's face will be exposed to a light source using blue light phototherapy machine between 15 to 20 minutes. The duration of each session will be approximately 20 minutes.
  Arms: BLP arm (Blue Light Phototherapy)
Device: Microcurrent therapy — Microcurrent therapy (Micro Current Electro-Device w/gloves and carrying case, SKU:DSE-X1008 Classic Spa Collection) The investigators will place one electrode in one of the regional areas of the lymph nodes or affected area (i.e. the forehead) and move the second electrode systematically from the affected area towards the stationary electrode. Once the entire affected area has been covered, the investigators will move the first electrode to another regional area of the lymph nodes or affected area and the process will be repeated. This will continue until all of the affected areas have been treated. The duration of each session will be approximately 45 minutes.
  Arms: MCT arm (Microcurrent Therapy)
Device: Combination of BLP and Microcurrent — Same devices as described above. At each session, participants will receive MCT portion as described in above followed by BLP portion as described above. These visits will last approximately 65 minutes.
  Arms: Combination of BLP and Microcurrent

SUMMARY:
Acne vulgaris is a multifactorial, highly prevalent dermatologic condition that results in visible lesions that can be quite disfiguring. Consequently, individuals with acne often suffer from a wide range of psychological manifestations. Although there is consensus that combination therapy is most effective in treating acne, researchers are constantly striving to develop new treatment. Microcurrent therapy (MCT) is a non-invasive modality that has successfully been used to promote wound healing and has been routinely used in aesthetics. Use of MCT alone or in combination with current successful treatment such as blue light phototherapy (BLP), may hold promise for acne treatment. The investigators propose to conduct a small randomized control trial to determine the safety and preliminary efficacy of a novel combination therapy to treat acne vulgaris. The investigators will recruit up to 60 males and females and randomly assign them to one of 3 arms: 1) BLP; 2) MCT; and combination therapy (BLP and MCT). The investigators will assess physiological parameters (number of acne lesions, amount of sebum produced, degree of acne severity) and psychosocial factors (dermatologic quality of life, social anxiety, depressive symptomatology, self-esteem). Participants will complete a baseline assessment prior to initiating treatment and a follow-up assessment at 4 weeks post termination of treatment. The investigators will conduct intermediary assessments at weeks 3 and 5 and 1 week post termination of the treatment. The investigators will use measures of central tendency to describe the sample and repeated measures analysis of variance to compute the main and interaction effects.

DETAILED DESCRIPTION:
Overview: The goal of this study is to conduct a small randomized control trial (RCT) to test the safety and preliminary efficacy of a novel combination therapy to treat acne vulgaris. The investigators will also explore the effects of the treatments on psychosocial factors (Dermatology Life Quality Index (DLQI), social anxiety, depressive symptomatology, and self-esteem). The RCT will have 3 arms: 1) FDA approved treatment: blue light phototherapy (BLP); 2) Microcurrent therapy (MCT); and 3) combination therapy (BLP + MCT). The main outcomes will be: 1) number of acne lesions; 2) amount of sebum produced, 3) degree of acne severity; and 4) improvement in dermatologic quality of life. The specific aims of the study are:

Aim 1: To explore the use of MCT to improve blood flow and lymphatic drainage and promote tissue repair in patients with acne vulgaris.

Aim 2: To examine the safety and preliminary efficacy of enhancing traditional blue light therapy treatment with microcurrent therapy (BLP + MCT) to promote faster healing in patients with acne vulgaris.

Aim 3: To determine if combination therapy is a more effective (fewer number of acne lesions, decreased amount of sebum produced, lesser degree of acne severity and greater improvement in dermatologic quality of life) for acne than either type of monotherapy.

Aim 4: To explore the effects of the three modalities on psychosocial factors (social anxiety, depressive symptomatology, and self-esteem).

The investigators will recruit up to 60 males and females and randomly assign them to one of 3 treatment arms (blue light phototherapy (BLP); microcurrent therapy (MCT); and combination therapy (BLP and MCT). All participants will complete a baseline assessment prior to initiating treatment one follow-up assessment at 4 weeks post termination of treatment. During the treatment phase, the investigators will conduct intermediary assessments to track the progression of the treatment over time at weeks 3 and 5 as well as 1 week post the termination of the treatment (week 6). The investigators will conduct both physiological and psychosocial assessments; the content of the intermediary assessment will be much less than the other 3 assessments to reduce participant data. The most comprehensive assessments will be conducted at baseline and one follow-up points and will consist of all of the physiological and psychosocial factors as well as demographic factors that will be collected exclusively at the baseline assessment. At the intermediary assessments, the investigators will collect the number of acne lesions, amount of sebum produced and dermatologic quality of life. Psychosocial data will be collected via computer-assisted self-interviews (CASI). Physiological data will be entered into the computer program by research staff.

Procedures for collecting psychosocial data: All assessments will be conducted using computer-assisted self-interviews (CASI). Participants will be assigned a unique study identification number (ID) that will be used to track data. Computer-assisted self-interviews are more effective than other tools for measuring sensitive and socially stigmatized behaviors. This mode of data collection eliminates interviewer bias, standardizes questionnaire administration, and reduces skip pattern errors. Using CASI, the participant responds to the questions using the computer keyboard or mouse. Selection of CASI for data collection decreases costs and error of entry, cleaning data, and publication lag, as well as enhances interviewer efficiency. The laptop computers the investigators use for data collection have been set up with two different log-in screens, one for participants and one for an administrator. The screen used by participants only contains the icon to access the CASI system. No other files appear or are available on this screen. The investigators access the CASI for participants by clicking the icon and filling in the assigned participant ID number (not participant name) completing all set up procedures. The investigator then provides a brief training on using the laptop and completing the CASI. As part of this training, the participant will complete a brief set of practice questions illustrative of the type of questions and the responses contained in the assessment. The investigator remains with the participant during the practice session to answer questions or to provide additional instructions. Participants will be encouraged to seek assistance, if needed, as they complete the interview. At this point, the interview starts and the participant completes the interview on their own. Once the participant completes the interview, he/she comes upon a screen instructing him/her to contact the investigators so that the file may be saved correctly.

Procedures for collecting physiological data: The investigators will conduct visual inspection of the affected areas and systematically count the number of acne lesions present on the face. At baseline and the follow-up assessment the investigators will also take high quality digital photographs of the affected areas that will be used to compute the degree of acne severity. The photographs will be identified exclusively by study ID and will be kept in a password protected file in a secure NSU computer. The Sebumeter® SM 815 sebum meter will be used to estimate the amount of sebum produced. The investigators will bring the mat tape of the meter in contact with the affected areas. This instrument uses a non-invasive probe placed on the affected area and the instrument then calculates the amount of sebum produced.

ELIGIBILITY:
Inclusion Criteria:

* Have mild to moderate facial acne
* Have Fitzpatrick skin type II-V
* Be able to understand written and/or spoken English
* Be able to provide written informed consent.

Exclusion Criteria:

* Have been treated with oral retinoids in the past 6 months
* Have been treated with oral antibiotic within the last 30 days
* Have received topical acne treatment (i.e. retinoids, antibiotics and anti-inﬂammatory agents or chemical peeling) within the last 30 days
* Pregnant or lactating
* Have history of photo-sensitive dermatitis
* Have previously received light therapy
* Taking oral contraceptive pills (OCP)
* Have pacemaker

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2014-10-30 (Actual); Primary Completion 2017-05-12 (Actual); Study Completion 2017-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Arutyunyan, M.S., Principal Investigator — Nova Southeastern University College of Osteopathic Medicine
Locations (2):
- United States (2):
  - NSU COM Division of Dermatology, General, Cosmetic Dermatology and Cutaneous Surgery, Fort Lauderdale, Florida
  - Hollywood Dermatology, Hollywood, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uhlenhake E, Yentzer BA, Feldman SR. Acne vulgaris and depression: a retrospective examination. J Cosmet Dermatol. 2010 Mar;9(1):59-63. doi: 10.1111/j.1473-2165.2010.00478.x. PMID 20367674
- [Background] Gollnick H, Cunliffe W, Berson D, Dreno B, Finlay A, Leyden JJ, Shalita AR, Thiboutot D; Global Alliance to Improve Outcomes in Acne. Management of acne: a report from a Global Alliance to Improve Outcomes in Acne. J Am Acad Dermatol. 2003 Jul;49(1 Suppl):S1-37. doi: 10.1067/mjd.2003.618. No abstract available. PMID 12833004
- [Background] Cunliffe WJ. The sebaceous gland and acne--40 years on. Dermatology. 1998;196(1):9-15. doi: 10.1159/000017859. No abstract available. PMID 9557218
- [Background] Gupta MA, Gupta AK. Depression and suicidal ideation in dermatology patients with acne, alopecia areata, atopic dermatitis and psoriasis. Br J Dermatol. 1998 Nov;139(5):846-50. doi: 10.1046/j.1365-2133.1998.02511.x. PMID 9892952
- [Background] Ashkenazi H, Malik Z, Harth Y, Nitzan Y. Eradication of Propionibacterium acnes by its endogenic porphyrins after illumination with high intensity blue light. FEMS Immunol Med Microbiol. 2003 Jan 21;35(1):17-24. doi: 10.1111/j.1574-695X.2003.tb00644.x. PMID 12589953
- [Background] Cheng N, Van Hoof H, Bockx E, Hoogmartens MJ, Mulier JC, De Dijcker FJ, Sansen WM, De Loecker W. The effects of electric currents on ATP generation, protein synthesis, and membrane transport of rat skin. Clin Orthop Relat Res. 1982 Nov-Dec;(171):264-72. PMID 7140077
- [Background] Bach S, Bilgrav K, Gottrup F, Jorgensen TE. The effect of electrical current on healing skin incision. An experimental study. Eur J Surg. 1991 Mar;157(3):171-4. PMID 1678624
- [Background] Carley PJ, Wainapel SF. Electrotherapy for acceleration of wound healing: low intensity direct current. Arch Phys Med Rehabil. 1985 Jul;66(7):443-6. PMID 3893385

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated and the PI has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Groups:
- MCT Arm (Microcurrent Therapy): In this arm participants will receive 5 MCT sessions 1 week intervals using MCT machine. The duration of each session will be approximately 45 minutes. The investigators will place one electrode in one of the regional areas of the lymph nodes or affected area (i.e. the forehead) and move the second electrode systematically from the affected area towards the stationary electrode. Once the entire affected area has been covered, the investigators will move the first electrode to another regional area of the lymph nodes or affected area and the process will be repeated. This will continue until all of the affected areas have been treated.
  Microcurrent therapy: The investigators will place one electrode in one of the regional areas of the lymph nodes or affected area (i.e. the forehead) and move the second electrode systematically from the affected area towards the statio
Period: Overall Study
Arm/Group | BLP Arm (Blue Light Phototherapy) | MCT Arm (Microcurrent Therapy) | Combination of BLP and Microcurrent
Started | 0 (The results cannot be evaluated because the sample size was so small. He had trouble recruiting) | 0 (The results cannot be evaluated because the sample size was so small. He had trouble recruiting) | 0 (The results cannot be evaluated because the sample size was so small. He had trouble recruiting)
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated and the PI has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Groups:
- Total: Total of all reporting groups
Arm/Group | BLP Arm (Blue Light Phototherapy) | MCT Arm (Microcurrent Therapy) | Combination of BLP and Microcurrent | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment
Have mild to moderate facial acne nd have Fitzpatrick skin type II-V

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Acne Lesions Over the Course of 9 Weeks
Description: The investigators will conduct a systematic count of acne lesions (papules and pustules) present in all of the affected areas of the face.
Time Frame: Weeks 1,3,5,6,9
Population: as for baseline characteristics
Groups:
- MCT Arm (Microcurrent Therapy): In this arm participants will receive 5 MCT sessions 1 week intervals using MCT machine. The duration of each session will be approx 45 minutes. The investigators will place one electrode in one of the regional areas of the lymph nodes or affected area and move the second electrode systematically from the affected area towards the stationary electrode. Once the entire affected area has been covered, the investigators will move the first electrode to another regional area of the lymph nodes or affected area and the process will be repeated. This will continue until all of the affected areas have been treated.
  Microcurrent therapy: Microcurrent therapy (Micro Current Electro-Device w/gloves and carrying case, SKU:DSE-X1008 Classic Spa Collection) The investigators will place one electrode in one of the regional areas of the lymph nodes or affected area (i.e. the forehead) and move the second electrode systematically from the affected area towards the statio
Arm/Group | BLP Arm (Blue Light Phototherapy) | MCT Arm (Microcurrent Therapy) | Combination of BLP and Microcurrent
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Change in the Amount of Sebum Produced Over the Course of 9 Weeks
Description: The investigators will use the Sebumeter® SM 815 manufactured by CK Electronic to estimate the amount of sebum. The measurement is based on grease spot photometry. The mat tape of the Sebumeter® SM 815 is brought into contact with facial skin. It becomes transparent in relation to the sebum on the surface of the measurement area. Then the tape is inserted into the aperture of the device and the transparency is measured by a photocell. The light transmission represents the sebum content.
Time Frame: Weeks 1,3,5,6,9
Population: as for baseline characteristics
Arm/Group | BLP Arm (Blue Light Phototherapy) | MCT Arm (Microcurrent Therapy) | Combination of BLP and Microcurrent
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Change in Acne Severity Over the Course of 9 Weeks
Description: The investigators will use the acne counts and the digital photographs of the affected areas to compute the acne severity level following the procedures established by Hayashi et al. (2008). The investigators will not print the digital photographs. The investigators will visually inspect the digital photographs and assign a preliminary severity score to each half of the face using the following classification guide: 0-5 papules and/pustules for mild acne; 6-20 for moderate acne, 21-50 for severe acne; and more than 50 for very severe. The investigators will examine each half of the face separately. The most severe classification obtained for either side of the face will be the assigned severity score.
Time Frame: Weeks 1 and 9
Population: as for baseline characteristics
Groups:
- MCT Arm (Microcurrent Therapy): In this arm participants will receive 5 MCT sessions 1 week intervals using MCT machine. The duration of each session will be approximately 45 minutes. The investigators will place one electrode in one of the regional areas of the lymph nodes or affected area and move the second electrode systematically from the affected area towards the stationary electrode. Once the entire affected area has been covered, the investigators will move the first electrode to another regional area of the lymph nodes or affected area and the process will be repeated. This will continue until all of the affected areas have been treated.
  Microcurrent therapy: Microcurrent therapy (Micro Current Electro-Device w/gloves and carrying case, SKU:DSE-X1008 Classic Spa Collection) The investigators will place one electrode in one of the regional areas of the lymph nodes or affected area (i.e. the forehead) and move the second electrode systematically from the affected area towards the statio
Arm/Group | BLP Arm (Blue Light Phototherapy) | MCT Arm (Microcurrent Therapy) | Combination of BLP and Microcurrent
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: Change in Dermatologic Quality of Life Over the Course of 9 Weeks
Description: The investigators will use the Dermatology Life Quality Index (DLQI) developed by A. Y. Finlay and G. K. Khan (1992), one of the most widely used, dermatologic specific quality of life measures in the published literature to assess quality of life. The DLQI consists of 10 Likert type items; 9 of these items have 4 response categories scored from 0 to 3 with "very much" being "3" to "not at all" being "0". Item 7 "Over the last week, has participant's skin prevented participant from working or studying" uses dichotomous responses; where "yes" is scored as a "3" and a "no" requires answering an additional sub-question, "Over the past week how much has participant's skin been a problem at work or studying". Responses for this sub-question range from "a lot" coded a "2", to "not at all" coded a "0." The DLQI is calculated by summing the response to each question; the maximum score is "30" and the minimum score is "0". The higher the score, the lower the dermatologic quality of life.
Time Frame: Weeks 1,3,5,6,9
Population: as for baseline characteristics
Arm/Group | BLP Arm (Blue Light Phototherapy) | MCT Arm (Microcurrent Therapy) | Combination of BLP and Microcurrent
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Change in Social Anxiety Score Over the Course of 9 Weeks
Description: Symptoms of social anxiety will be assessed using the Liebowitz Social Anxiety Scale (Liebowitz, 1987), one of the most widely used scales to measure social anxiety. It consists of 24 items designed to assess fear and avoidance in different situations that are likely to produce social anxiety such as going to a party or speaking in public. For each situation, participants are first asked to state how fearful or anxious they feel in that situation using a Likert scale that ranges from "none" (0) to "severe" (3). Then they are asked to state how often they avoid that same situation using a Likert scale that ranges from "never" (0) to "usually" (3). Responses are summed to create an overall anxiety score.
Time Frame: Weeks 1 and 9
Population: as for baseline characteristics
Arm/Group | BLP Arm (Blue Light Phototherapy) | MCT Arm (Microcurrent Therapy) | Combination of BLP and Microcurrent
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Change in Depressive Symptomatology Score Over the Course of 9 Weeks
Description: The investigators will assess depressive symptomatology using the Hospital Anxiety and Depression Scale (HADS) (Zigmond and Snaith 1983), one of the most widely used screening tools to identify symptoms of depression, anxiety and emotional distress amongst patients being treated for a variety of clinical problems. It consists of 14 items, 7 of which assess generalized symptoms of anxiety and the remaining 7 assess depressive symptomatology. Although the specific wording of the item responses vary in accordance to the item, all responses are coded using a Likert format ranging from "0" to "3" where the most positive response is coded a "0" and the most negative response a "3". The maximum score for each subscale is 21; higher scores are reflective of more symptoms of anxiety or depression.
Time Frame: Weeks 1 and 9
Population: as for baseline characteristics
Arm/Group | BLP Arm (Blue Light Phototherapy) | MCT Arm (Microcurrent Therapy) | Combination of BLP and Microcurrent
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Change of Self-esteem Score Over the Course of 9 Weeks
Description: Self-esteem will be assessed using the Rosenberg Self-Esteem Scale, one of the most widely-used self-esteem measures in social science research. It consists of ten items designed to assess respondent's self-satisfaction, self-respect and other general feelings about himself/herself. The response format is a four point Likert scale ranging from "strongly agree" to "strongly disagree". For items 1, 2, 4, 6, 7: Strongly Agree=3, Agree=2, Disagree=1, and Strongly Disagree=0. For items 3, 5, 8, 9, 10: Strongly Agree=0, Agree=1, Disagree=2, and Strongly Disagree=3. The scale ranges from 0-30, higher scores indicating higher self-esteem.
Time Frame: Weeks 1 and 9
Population: as for baseline characteristics
Arm/Group | BLP Arm (Blue Light Phototherapy) | MCT Arm (Microcurrent Therapy) | Combination of BLP and Microcurrent
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 years
Description: The study was terminated and the PI has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Arm/Group | BLP Arm (Blue Light Phototherapy) | MCT Arm (Microcurrent Therapy) | Combination of BLP and Microcurrent
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2014-08-29): https://cdn.clinicaltrials.gov/large-docs/94/NCT02431494/Prot_SAP_ICF_000.pdf